CLINICAL TRIAL: NCT06907628
Title: A Phase Ⅰ, Open Label, Multicenter Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of SHR-3792 in Patients With Advanced Solid Tumors
Brief Title: A Trial of SHR-3792 Injection in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-3792-101
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-3792 Injection Group (Experimental)
  Interventions: Drug: SHR-3792 Injection

INTERVENTIONS:
Drug: SHR-3792 Injection — SHR-3792 injection.

SUMMARY:
The study is being conducted to evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of SHR-3792 injection monotherapy for patients with advanced solid tumors, and to explore the reasonable dosage of SHR-3792 injection monotherapy for patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with ability to understand and voluntarily agree to participate by giving written informed consent form for the study.
2. Patients with unresectable recurrent or metastatic solid tumors.
3. There is at least one lesion that could be measured.
4. An Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 1.
5. Adequate organ functions as defined.
6. Life expectancy ≥ 3 months.

Exclusion Criteria:

1. Patients with known active central nervous system (CNS) metastases.
2. Subjects with other malignancy in five years before the first dose.
3. Patients with tumor-related pain that cannot be controlled as determined.
4. Patients with serious cardiovascular and cerebrovascular diseases.
5. Uncontrollable third-space effusion, such as pleural effusion, pericardial effusion or peritoneal effusion.
6. Patients with severe infections.
7. History of immunodeficiency.
8. History of autoimmune diseases.
9. Active infection.
10. Pregnant or nursing women.
11. Known history of serious allergic reactions to the investigational product or its main ingredients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | From the first dose of study medication up to 21 days.
Recommended phase Ⅱ dose (RP2D) | From the first dose of study medication up to 21 days.
Incidence of dose limited toxicity (DLT) | From the first dose of study medication up to 21 days.
Adverse events (AEs) | Up to 24 weeks.
Serious adverse events (SAEs) | Up to 24 weeks.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong First Medical University Affiliated Cancer Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided